CLINICAL TRIAL: NCT03108989
Title: Comparison the Postoperative Quality of Recovery Between Neostigmine and Sugammadex in Elderly Patients Undergoing Trans Pars Plana Vitrectomy With General Anesthesia -Randomized Controlled Trial-
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2015-0641
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Elderly Patients Undergoing Trans Pars Plana Vitrectomy With General Anesthesia
MeSH Terms: interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex group (Experimental): After the end of surgery, sugammadex of 2 mg/kg will be administered to reverse neuromuscular blockade.
  Interventions: Drug: Sugammadex
- Neostigmine group (Active Comparator): After the end of surgery, neostigmine will be administered to reverse neuromuscular blockade.
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — After the end of surgery, sugammadex of 2 mg/kg will be administered to reverse neuromuscular blockade.
  Arms: Sugammadex group
Drug: Neostigmine — After the end of surgery, neostigmine will be administered to reverse neuromuscular blockade.
  Arms: Neostigmine group

SUMMARY:
Sugammadex has been approved as the first targeted reversal binding agent providing predictable and complete reversal of neuromuscular blockade induced by rocuronium or vecuronium, and achieving so with a favourable safety profile.

Its benefits over traditional acetylcholinesterase inhibitors have been widely demonstrated in many studies. The scope of such studies has been mostly related to the efficacy of NMB reversal and safety. However, the clinical use of sugammadex led some anaesthesiologists to observe that following the use of this agent, patients seemed to recover consciousness faster and look like they were feeling better. To present, there is little information on the effect of sugammadex on awakening from anaesthesia.

The quality of postoperative recovery focused around patient-oriented endpoints has raised new interest as a measure of the quality of anaesthesia and a target towards which improvement can be directed.

On the other hand, there is no single prospective study performed to address a possible effect of sugammadex on recovery from anaesthesia.

The objective of this study was to compare the effect of sugammadex and neostigmine on the quality of postoperative recovery using the PQRS in elderly patients undergoing trans pars plana vitrectomy with general anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged over 60 years who are scheduled for trans pars plana vitrectomy with general anesthesia

Exclusion Criteria:

* Neuromuscular disease
* History of malignant hyperthermia
* Significant renal or hepatic dysfunction
* Allergy to sugammadex or rocuronium
* BMI > 30kg/m2
* History of medication which affect neuromuscular blocker such as anti-convulsants, magnesium

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-07-25 (Actual); Study Completion 2017-07-25 (Actual)

PRIMARY OUTCOMES:
physiological domain of PQRS recovery | at 40 min after the end of surgery
  The primary objective of the study was to assess the physiological domain of PQRS recovery from anesthesia for patients treated with neostigmine and those given sugammadex at 40 min after the end of surgery. Recovery was defined as return (or improvement from) baseline values.

SECONDARY OUTCOMES:
overall PQRS recovery and recovery in the different domains of the PQRS | The secondary objective of the study was to compare the overall PQRS recovery and recovery in the different domains of the PQRS between neostigmine and sugammadex treated patients at 15 min , 40 min , 1 day after the end of surgery.
  at 15 min, 40 min , 1 day after the end of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim NY, Koh JC, Lee KY, Kim SS, Hong JH, Nam HJ, Bai SJ. Influence of reversal of neuromuscular blockade with sugammadex or neostigmine on postoperative quality of recovery following a single bolus dose of rocuronium: A prospective, randomized, double-blinded, controlled study. J Clin Anesth. 2019 Nov;57:97-102. doi: 10.1016/j.jclinane.2019.02.014. Epub 2019 Mar 30. PMID 30939422